CLINICAL TRIAL: NCT00367003
Title: Deep Brain Stimulation for Treatment Resistant Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Dana Foundation (Other)
Responsible Party: Principal Investigator, Patricio Riva Posse, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024883
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression, Unipolar, Bipolar-II, DBS, Imaging
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Participants with treatment resistant depression will have a device implanted for deep brain stimulation.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — The deep brain stimulation system (consisting of a lead, extension wire, and implanted pulse generator) will be surgically implanted to stimulate the targeted area of the brain. Stimulation will be turned off for 4 weeks following implantation, then participants will use brain stimulation for 6 months. Participants will also take part in Behavioral Activation therapy during the 6 months of active stimulation. Participants will be followed for 10 years, or until the DBS device has been FDA approved, with adjustments made to the stimulator and medications as necessary.

SUMMARY:
The purpose of this study is to test the safety, efficacy and mechanism of action of subgenual cingulate (Cg25) deep brain stimulation (DBS) for major depression in patients who have not responded to prior antidepressant treatments. Participation in the study will continue for ten years or until the device receives FDA approval for depression. Forty (40) patients will be enrolled in this study.

DETAILED DESCRIPTION:
Major Depression is one of the most common and costly of all psychiatric disorders. While depression can be effectively treated in the majority of patients by either medication or some form of evidence-based psychotherapy, up to 20% of patients fail to respond to standard interventions. For these patients, trial-and-error combinations of multiple medications and electroconvulsive therapy are often required. For patients who remain severely depressed despite these aggressive approaches, new strategies are needed.

Converging clinical, biochemical, neuroimaging, and post-mortem data suggest depression is unlikely to be a disease of a single brain region or neurotransmitter system. Rather, it is now generally viewed as a systems-level disorder affecting integrated pathways linking select cortical, subcortical and limbic sites and their related neurotransmitter and molecular mediators. Treatments for depression can be viewed within a limbic-cortical system framework, where different modes of treatment modulate specific regional targets, resulting in a variety of complementary, adaptive chemical and molecular changes that re-establish a normal mood state. Functional neuroimaging studies have played a critical role in characterizing these limbic-cortical pathways. Previous studies have demonstrated consistent involvement of the subgenual cingulate (Cg25) in both acute sadness and antidepressant treatment effects, suggesting a critical role for this region in modulating negative mood states.

This study will test whether high frequency deep brain stimulation of the subgenual cingulate white matter (Cg25-DBS) is a safe and efficacious antidepressant treatment in forty patients with treatment resistant depression, and to investigate potential mechanisms of action of this intervention.

ELIGIBILITY:
Inclusion criteria:

* Ability to provide written informed consent.
* Current Major Depressive Episode (MDE), secondary to either Major Depressive Disorder or Bipolar Disorder (I, II or NOS), diagnosed by structured clinical interview for Diagnostic and Statistical Manual of Mental Disorders-IV-text revision (DSM-IV-TR).
* Current MDE at least two years duration OR a history of more than 4 lifetime depressive episodes.
* Minimum score at study entry of 20 on the 17-item Hamilton Depression Rating Scale (HDRS-17).
* Average pre-operative HDRS-17 score of 20 or greater (averaged over four weekly pre-surgical evaluations during the four weeks prior to surgery) and an average pre-operative HDRS-17 score no more than 30% lower than the baseline screening HDRS-17 score.
* A maximum Global Assessment of Functioning of 50.
* Treatment-resistant depression defined as:

  * Failure to respond to a minimum of four different antidepressant treatments, including at least three medications from at least three different classes, evidence-based psychotherapy or electroconvulsive therapy (ECT) administered at adequate doses and duration during the current episode.
  * Failure or intolerance of an adequate course of electroconvulsive therapy (ECT) during any episode (confirmed by medical records), or refusal of ECT due to a reason considered to be valid by the study psychiatrist.
* A patient may remain on psychotropic medications during this study. However, doses must remain stable during the 4 weeks prior to surgery, the four weeks post-operatively, and the 24 weeks open stimulation phase. Medications will be changed only if intolerable side effects clearly attributable to the medications develop.
* All patients must have an established outpatient psychiatrist and be willing to sign a written release to allow study investigators to give and receive information from this psychiatrist.

Exclusion criteria:

* Inability to tolerate general anesthesia.
* Significant cerebrovascular risk factors or a previous stroke, documented major head trauma or neurodegenerative disorder.
* Other currently active clinically significant Axis I psychiatric diagnosis including schizophrenia, panic disorder, obsessive-compulsive disorder, generalized anxiety disorder or post-traumatic stress disorder. Patients with severe Axis II personality disorders will also be excluded if the personality disorder is likely to interfere with cooperation and adherence to the study protocol.
* Current psychotic symptoms.
* Evidence of global cognitive impairment.
* Substance abuse or dependence not in full sustained remission (i.e., not active for at least one year).
* Active suicidal ideation with intent; suicide attempt within the last six months; more than three suicide attempts within the last two years.
* Pregnancy or plan to become pregnant during the study period.
* General contraindications for DBS surgery (cardiac pacemaker/defibrillator or other implanted devices).
* Inability or unwillingness to comply with long-term follow-up.
* History of intolerance to neural stimulation of any area of the body.
* Participation in another drug, device or biologics trial within the preceding 30 days.
* Conditions requiring repeated MRI scans.
* Conditions requiring diathermy.
* Conditions requiring anticoagulant medication.
* Terminal illness associated with expected survival of <12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-09; Primary Completion 2014-01-02 (Actual); Study Completion 2029-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Riva Posse, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Riva-Posse P, Crowell AL, Wright K, Waters AC, Choi K, Garlow SJ, Holtzheimer PE, Gross RE, Mayberg HS. Rapid Antidepressant Effects of Deep Brain Stimulation and Their Relation to Surgical Protocol. Biol Psychiatry. 2020 Oct 15;88(8):e37-e39. doi: 10.1016/j.biopsych.2020.03.017. Epub 2020 May 14. No abstract available. PMID 32418613
- [Result] Crowell AL, Riva-Posse P, Holtzheimer PE, Garlow SJ, Kelley ME, Gross RE, Denison L, Quinn S, Mayberg HS. Long-Term Outcomes of Subcallosal Cingulate Deep Brain Stimulation for Treatment-Resistant Depression. Am J Psychiatry. 2019 Nov 1;176(11):949-956. doi: 10.1176/appi.ajp.2019.18121427. Epub 2019 Oct 4. PMID 31581800
- [Result] Riva-Posse P, Choi KS, Holtzheimer PE, Crowell AL, Garlow SJ, Rajendra JK, McIntyre CC, Gross RE, Mayberg HS. A connectomic approach for subcallosal cingulate deep brain stimulation surgery: prospective targeting in treatment-resistant depression. Mol Psychiatry. 2018 Apr;23(4):843-849. doi: 10.1038/mp.2017.59. Epub 2017 Apr 11. PMID 28397839
- [Result] Holtzheimer PE, Kelley ME, Gross RE, Filkowski MM, Garlow SJ, Barrocas A, Wint D, Craighead MC, Kozarsky J, Chismar R, Moreines JL, Mewes K, Posse PR, Gutman DA, Mayberg HS. Subcallosal cingulate deep brain stimulation for treatment-resistant unipolar and bipolar depression. Arch Gen Psychiatry. 2012 Feb;69(2):150-8. doi: 10.1001/archgenpsychiatry.2011.1456. Epub 2012 Jan 2. PMID 22213770
- [Result] Riva-Posse P, Choi KS, Holtzheimer PE, McIntyre CC, Gross RE, Chaturvedi A, Crowell AL, Garlow SJ, Rajendra JK, Mayberg HS. Defining critical white matter pathways mediating successful subcallosal cingulate deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2014 Dec 15;76(12):963-9. doi: 10.1016/j.biopsych.2014.03.029. Epub 2014 Apr 13. PMID 24832866
- [Derived] Filkowski MM, Mayberg HS, Holtzheimer PE. Considering Eligibility for Studies of Deep Brain Stimulation for Treatment-Resistant Depression: Insights From a Clinical Trial in Unipolar and Bipolar Depression. J ECT. 2016 Jun;32(2):122-6. doi: 10.1097/YCT.0000000000000281. PMID 26479487
- [Derived] Riva-Posse P, Holtzheimer PE, Garlow SJ, Mayberg HS. Practical considerations in the development and refinement of subcallosal cingulate white matter deep brain stimulation for treatment-resistant depression. World Neurosurg. 2013 Sep-Oct;80(3-4):S27.e25-34. doi: 10.1016/j.wneu.2012.11.074. Epub 2012 Dec 13. PMID 23246630
- [Derived] Fisher CE, Dunn LB, Christopher PP, Holtzheimer PE, Leykin Y, Mayberg HS, Lisanby SH, Appelbaum PS. The ethics of research on deep brain stimulation for depression: decisional capacity and therapeutic misconception. Ann N Y Acad Sci. 2012 Aug;1265:69-79. doi: 10.1111/j.1749-6632.2012.06596.x. Epub 2012 Jul 19. PMID 22812719
- [Derived] Christopher PP, Leykin Y, Appelbaum PS, Holtzheimer PE 3rd, Mayberg HS, Dunn LB. Enrolling in deep brain stimulation research for depression: influences on potential subjects' decision making. Depress Anxiety. 2012 Feb;29(2):139-46. doi: 10.1002/da.20916. Epub 2011 Nov 17. PMID 22095837
- [Derived] Holtzheimer PE 3rd, Mayberg HS. Deep brain stimulation for treatment-resistant depression. Am J Psychiatry. 2010 Dec;167(12):1437-44. doi: 10.1176/appi.ajp.2010.10010141. No abstract available. PMID 21131410

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 participants were consented but only 28 participants underwent Subcallosal Cingulate Deep Brain Stimulation (DBS) between January 2007 and June 2013.
Period: Overall Study
Arm/Group | Deep Brain Stimulation
Started | 37
Completed | 28
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: 28 participants underwent Subcallosal Cingulate Deep Brain Stimulation between January 2007 and June 2013.
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
  Not reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 28
Hamilton Depression Rating Scale Score [Mean (Standard Deviation); unit: score on a scale] | 23.6 (2.9)
Number of medications at time of implantation surgery [Mean (Standard Deviation); unit: number of medications] | 3.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Rating Scale-17 Score
Description: The Hamilton Depression Rating Scale (HDRS-17) contains 17 items that are scored from 0 to 2, 3, or 4, where 0 is lack of difficulty and the highest number for an item is the most extreme difficulty. Total scores range from 0 to 53 and higher scores indicate greater depression. For this study, a response to treatment will be defined as a decrease in the HDRS-17 score of 50% or greater from the average pre-surgical baseline.
Time Frame: Baseline, Week 24 post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deep Brain Stimulation
Number analyzed (Participants) | 28
score on a scale
  Baseline | 23.6 (2.9)
  Week 24 post-intervention | 11.66 (2.6)

ADVERSE EVENTS:
Time Frame: Data for Adverse Events and Severe Adverse Events was collected during follow up time of the Primary Outcome (up to 24 weeks post intervention).
Arm/Group | Deep Brain Stimulation
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 6/28
Other Adverse Events (participants affected / at risk) | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation (N=28)
Infection (General disorders) | 2 (2)
Syncope (General disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Cap Erosion with dehissence of suture line (Injury, poisoning and procedural complications) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Axiety requiring hospitalization (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deep Brain Stimulation (N=28)
Paresthesia (Nervous system disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Worsening Depression (Psychiatric disorders) | 3 (3)
Weakness (General disorders) | 1 (1)
DBS system revision as a result of dislodgement (Injury, poisoning and procedural complications) | 1 (1)
Sinus Infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Car accident (Injury, poisoning and procedural complications) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT00367003/Prot_SAP_000.pdf